CLINICAL TRIAL: NCT00256464
Title: Evaluation of a Multi-Component Yoga Intervention as Adjunct to Psychiatric Treatment for Vietnam Veterans With Posttraumatic Stress Disorder (PTSD): A Randomized Controlled Trial (RCT).
Brief Title: Evaluation of a MCYI as Adjunct to Psychiatric Treatment for Vietnam Veterans With PTSD - RCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Queensland (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: MCYI-PTSD
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-08

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

INTERVENTIONS:
Behavioral: Multi-component Yoga Intervention

SUMMARY:
The principal aim of this project is to conduct a Randomized Controlled Trial (RCT) to examine whether adding a twelve-session Multi-Component Yoga Intervention (MCYI) to the treatment regimen of Australian Vietnam Veterans suffering chronic Posttraumatic Stress Disorder (PTSD) leads to a significantly greater clinical improvement than conventional psychiatric treatment alone. Include 12 sessions with each session 3 hours duration- 4 days per week for 3 weeks i.e. total of 36 hours. The Multi-Component Yoga Intervention (MCYI) consisting of specific poses, breathing techniques, information about yoga techniques and practices, group processes, psychoeducation, relaxation procedures and meditation techniques in Vietnam War Veterans with chronic Posttraumatic Stress Disorder (PTSD) resistant to treatment has been developed. This project aims to evaluate MCYI through RCT method.

It is hypothesised that Yoga augmentation will lead to: (1) reduced symptoms of PTSD and Depression; and (2) reduced alcohol intake. A secondary aim of the proposed RCT is to evaluate putative mediating variables. Benefits include that it is low cost and easy to apply. Done at home, non threatening and additional to standard psychiatric treatment for PTSD.

DETAILED DESCRIPTION:
The principal aim of this project is to conduct a Randomized Controlled Trial (RCT) to examine whether adding a twelve-session Multi-Component Yoga Intervention (MCYI) to the treatment regimen of Australian Vietnam Veterans suffering chronic Posttraumatic Stress Disorder (PTSD) leads to a significantly greater clinical improvement than conventional psychiatric treatment alone. Include 12 sessions with each session 3 hours duration- 4 days per week for 3 weeks i.e. total of 36 hours. The Multi-Component Yoga Intervention (MCYI) consisting of specific poses, breathing techniques, information about yoga techniques and practices, group processes, psychoeducation, relaxation procedures and meditation techniques in Vietnam War Veterans with chronic Posttraumatic Stress Disorder (PTSD) resistant to treatment has been developed. This project aims to evaluate MCYI through RCT method.

It is hypothesised that Yoga augmentation will lead to: (1) reduced symptoms of PTSD and Depression; and (2) reduced alcohol intake. A secondary aim of the proposed RCT is to evaluate putative mediating variables. Benefits include that it is low cost and easy to apply. Done at home, non threatening and additional to standard psychiatric treatment for PTSD.

A comparable method with a different emphasis is currently the subject of a United States grant application by another group to formally test American War Veterans from Afghanistan and Iraq. The chief investigators (Assistant Professor Gerbarg and Associate Professor Brown) are collaborating with The Bay Pines Veterans Administration Medical Center in Florida to develop a study utilising a specific Yoga breathing technique called Sudarshan Kriya Yoga (SKY) for treatment of American veterans returning from Afghanistan and Iraq. Elements of this method have been widely tested on individuals suffering with Acute Stress Disorder and Posttraumatic Stress Disorder (Gerbarg and Brown 2005 Direct communication) and have been reported to have relieved posttraumatic stress disorder (PTSD) in large groups of people affected by mass disasters such as: war (Kosovo, Bosnia, Iraq and Sudan) (Biswas 2004; Joseph 2004; Luedemann 2004); terrorism (New York City 9/11) (Anonymous 2001b), (Kashmir, India, Israel); and natural disasters (Gujurat earthquake, Iran flood and the Asian Tsunami) (Gujurat earthquake, 2000) (Anonymous 2001a). Pilot studies conducted by the Principal Investigator using similar techniques showed positive health results for Vietnam Veterans with PTSD in Australia (Carter and Byrne 2004).

(Kessler, Sonnega et al. 1995) studied the disabling effect of PTSD in their NCS study and conclude that PTSD and Major Depression are the two most substantial causes of burden of disease by psychological disorder. The Australian national epidemiology study (Creamer, Burgess et al. 2001) support this in analysis of work days lost per month (2.8 days per month.

Generally, evidence from a well-designed Random Controlled Trial (RCT) is accepted as having a high level of strength for efficacy. From the literature review, none of the outcome studies investigating the efficacy of yoga treatment for PTSD have been conducted by using RCT design. Most of the studies lack treatment control subjects and rely on data from only one program. Thus, it is expected the Multi-Component Yoga Intervention (MCYI) will be the first RCT study conducted internationally and will contribute significantly to the field of mental health and psychiatry.

However, although a randomized clinical trial has been performed for depression with good effect (Janakiramaiah, Gangadhar et al. 2000), there are as yet no randomized clinical trials testing the efficacy of a yoga intervention for Posttraumatic Stress Disorder in Vietnam Veterans. Accordingly, it is proposed to apply a Multi-Component Yoga Intervention (MCYI) for a group of Australian Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of PTSD DSM IV for a minimum of 12 months prior to screening meeting Mini Plus
* Satisfy CAPS test for PTSD having all criterions
* Alcohol Audit with a score of 8 or less in dependence
* An absence of suicidal intent, organic brain disease, absence of present psychosis identified

Exclusion Criteria:

* History of psychosis
* Subject with greater than 20% reduction in their CAPS 2 score between screening and baseline
* Those who are acutely suicidal
* Current substance dependence or abuse exept for alcohol
* Subject requiring electro convulsive therapy or who have had recent ECT which may cause interference with cognitive function.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-06; Study Completion 2008-01

PRIMARY OUTCOMES:
Decreased symptoms of posttraumatic stress disorder
Decreased symptoms of comorbid conditions of depression and alcohol dependence

CONTACTS AND LOCATIONS:
Overall Officials: Janis J Carter, MBBS FRANZCP, Principal Investigator — The University of Queensland

REFERENCES:
- See also: History of previous trials — http://www.therapywithyoga.com